CLINICAL TRIAL: NCT06734091
Title: Rapid Processing and Immunohistochemistry Method for Optimising Diagnosis Time in Solid Organ Donors With Suspected Malignancy
Brief Title: Rapid Processing and Immunohistochemistry Method for Optimising Diagnosis Time in Solid Organ Donors, Suspected Malignancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: donorEXT_2022; RC 2022-2024 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-12-01; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Donors; Organ Donor; Organ Transplants
Keywords: Transplants

STUDY DESIGN:
Intervention Model Description: Donors tissue will be send to Pathological Anatomy to perform intraoperative examination according to standard of care procedures and to perform intraoperative examination according to experimental methods (with possible immunohistochemistry).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donors undergoing intraoperative examination (Experimental): Donors undergoing intraoperative extemporaneous examination to define the oncological risk of donation during the study period
  Interventions: Diagnostic Test: PrestoCHILL

INTERVENTIONS:
Diagnostic Test: PrestoCHILL — PrestoCHILL (Milestone Medical Technologies, Inc.MI 49009, USA)which by reducing the tissue freezing time to less than 60 seconds should eliminate freezing artefacts and improve the quality of sections for morphological and IHC examination. In selected cases and according to the diagnostic algorithm required for the diagnosis of specific neoplasms, rapid IHC analysis will be performed with the Benchmark ULTRA® immunostainer (Ventana Medical Systems), which is already in place to confirm or exclude the suspected neoplasm, as well as to confirm the histotype. For the latter purpose, commercially available antibody panels for routine examinations will be used (Ventana/Roche,Ventana Medical Systems, USA).

SUMMARY:
Comparison of the diagnostic yield of intra-operative histological analysis of donor tissue with suspected neoplasia performed with the standard method versus the experimental method, which involves optimisation of sample freezing and analysis with the IHC fast track procedure

DETAILED DESCRIPTION:
Optimisation of frozen material can be achieved with specific tools that improve the quality of freezing and the cutting of histological sections, allowing a lower incidence of artefacts, with better histological definition. These instruments would also allow the execution of automated IHC protocols, with increased diagnostic sensitivity and specificity and better risk stratification for donors with malignancy. All this should lead to an increase in the donor pool with better oncological risk stratification and, consequently, increase the number of organs to be allocated, making it possible to respond more promptly to the great demand for organs needed for transplantation.

Moreover, not only would the certain exclusion of a neoplasm allow the use of donors who would otherwise have been considered to be at unacceptable risk and therefore excluded from the donor process, but a more precise diagnosis of the neoplasm (where present) would allow the second opinion to stratify the risk more accurately, with a more rational use of organs.

All organ donors who request extemporaneous intraoperative examinations to define the oncological risk of donation during the study period will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Organ donors (legally dead by brain or cardiac death) with suspected neoplasia.
* Sending organs/tissues of all types and locations for extemporaneous examination request

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of intraoperative histological analysis | Up to 20 months
  comparison of the diagnostic yield of intra-operative histological analysis of donor tissue with suspected neoplasia performed with the standard method versus the experimental method, which involves optimisation of sample freezing and analysis with the IHC fast track procedure.
  Increase in the number of donors used and the number of grafts (liver and kidneys, but also heart, lungs and 'bankable' tissues such as bones, vascular segments and corneas) that could be recovered and then used for transplantation due to better risk stratification of donors with malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Malvi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No